CLINICAL TRIAL: NCT06724250
Title: Biofeedback Versus Botox Injection in Treatment of Dyssynergic Defecation (Randomized Controlled Trial)
Brief Title: Biofeedback Therapy Versus Botox Injection in Treatment of Dyssynergic Defecation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.23.090.2539
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Obstructed Defaecation Syndrome
MeSH Terms: interventions — Biofeedback, Psychology; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biofeedback therapy group (Active Comparator): Patients with dyssynergic defecation underwent biofeedback training program in the form of six sessions over one month
  Interventions: Device: Biofeedback therapy
- Botox injection group (Active Comparator): Participants in this group received 100 international unit of botulinum toxin type A that was injected injections into the puborectalis muscle to alleviate dyssynergic defecation by reducing muscle overactivity and improving coordination.
  Interventions: Drug: Botulinum Toxin A (Botox )

INTERVENTIONS:
Device: Biofeedback therapy — Biofeedback therapy involves the use of specialized equipment to provide real-time feedback on pelvic floor muscle activity. Participants are trained to improve muscle coordination and relaxation through guided exercises, targeting the resolution of dyssynergic defecation.
  Arms: Biofeedback therapy group
Drug: Botulinum Toxin A (Botox ) — Botulinum toxin is injected into the pelvic floor muscles to reduce muscle overactivity and improve coordination, aiming to relieve symptoms of dyssynergic defecation.
  Arms: Botox injection group

SUMMARY:
assessment the Improvement symptoms of obstructed defecation after biofeedback training versus botulinum toxin injection

DETAILED DESCRIPTION:
This is a randomized controlled trial including 78 patients diagnosed with obstructed defecation syndrome confirmed by detailed history talking, full clinical examination, anorectal manometry and defecography.

Included patients divided into two equal groups: first group ( biofeedback therapy group) patients recieved biofeedback therapy for six sessions over one month, the second group:( botulinum toxin group) received botulinum toxin injection 100 IU in buborectalis muscle.

The primary outcome is improvement of symptoms after one year

ELIGIBILITY:
Inclusion Criteria:

* patients of both genders
* age of 18 years or older
* fulfillment of the Rome 3 constipation criteria for the past 3 months, symptom onset as a maximum six months prior to diagnosis, patients suffer from prolonged, incomplete and challenging evacuation

Exclusion Criteria:

* Anismus cases with secondary reason for constipation
* patients who undergone anorectal surgery Patients with colonic inertia
* conditions that make biofeedback training impossible
* cases with primary illness causing constipation as hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms of constipation for one year follow up | One year
  * Follow-up was conducted for about 1 year as regard the improvement in bowel habits.
  * Patients was asked to fill up a symptom questionnaire (Wexner constipation score with a maximum score of 30 and a minimum of 0) following the therapeutic procedure The wexner constipation score : include 8-item questionnaire about bowel movements frequency, anal pain during evacuation, abdominal pain, incomplete evacuation, time taken for evacuation per attempt, number of attempts for a successful bowel movement in the previous 24 hours, type of assistance for defecation, and duration of constipation. All items are scored from 0 to 4 except for the "type of assistance for defecation," which is scored from 0 to 2.The clinical improvement was chosen when there was decrease in the score.

SECONDARY OUTCOMES:
Improvement of pain for one year follow up | One year
  Pain improvement on the visual analogue scale is from 0 to 10, where 0 means no pain and 10 means the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code